CLINICAL TRIAL: NCT03324282
Title: Gemcitabine-cisplatin Plus Avelumab or Gemcitabine-cisplatin as First-line Treatment of Patients With Locally Advanced or Metastatic Urothelial Bladder Carcinoma (GCISAVE)
Brief Title: First-line Gemcitabine/Cisplatin +/- Avelumab in Locally Advanced or Metastatic Bladder Carcinoma
Acronym: GCISAVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: ANSM's refusal to validate ATU requests for avelumab in bladder cancer, Decrease in recruitment, Most investigators would like to offer avelumab for maintenance, Absence of benefit to the chemo-immuno combination (pembro+gem-platinum) in phase III
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2016/33
Record Dates: First submitted 2017-10-19; First posted 2017-10-27 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Bladder Carcinoma
Keywords: Anti PD1; Bladder carcinoma; Chemotherapy; Immunological monitoring
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: GC + avelumab group (Experimental)
  Interventions: Drug: Avelumab; Drug: GC
- Arm B: GC group (Active Comparator)
  Interventions: Drug: GC

INTERVENTIONS:
Drug: Avelumab — Combination of Gemcitabin-Cisplatin and avelumab given for 6 cycles (each cycle is 21 days)
  Arms: Arm A: GC + avelumab group
Drug: GC — Combination of Gemcitabin-Cisplatin given for 6 cycles (each cycle is 21 days)

SUMMARY:
This study will assess efficacy (based on response rate) and safety (based on grade ≥ 3 severe adverse effects) of the combination Gemcitabine Cisplatin (GC) + anti-PD-L1 (avelumab) in first-line treatment for locally advanced or metastatic urothelial bladder cancer patients, after 6 cycles of treatment (or at 18 weeks if less than 6 cycles have been given, or earlier if a second line treatment is needed, before this new anticancer treatment has been started).

DETAILED DESCRIPTION:
Recent results in cancer research highlight the importance of immune checkpoints in the control of immune response and provide access to molecules interfering with the inhibited immune response during the development of cancer. Drugs targeted against CTLA-4, PD-1 or PD-L1 have shown efficacy in various tumor types. In locally advanced or metastatic urothelial bladder cancer (MBC), the standard first-line treatment is the association of Gemcitabine and Cisplatin (GC). Objective responses and prolonged objective responses have been reported with monoclonal antibodies against PD-1 or PD-L1 in MBC patients after failure of chemotherapy. Avelumab is an investigational fully human anti-PD-L1 IgG1 monoclonal antibody. Avelumab treatment did not show unexpected cross-toxicity with chemotherapy when studied in phase I / II in patients with different tumor types. So the combination at full doses of GC and avelumab seems appropriate.

The experimental treatment is a combination of GC and avelumab given for 6 cycles. The duration of each cycle is 3 weeks (Gemcitabine: dose of 1000 mg/m2 as an intravenous infusion over 30 minutes on Days 1 and 8 of each 21-day cycle; Cisplatin: dose of 70 mg/m2 as a slow intravenous infusion over 2 to 4 hours on Day 1 of each 21-day cycle; Avelumab: 10 mg/kg body weight administered Iv once every 3 weeks).

Patients who have received all scheduled treatments and whose disease has not progressed at the end of treatment will enter into disease follow-up. During this follow-up period, patients will have disease and safety assessments performed every 3 months. Patients will remain in follow-up for up to 1 year from last dose of treatment and will have survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent;
2. Male or female, age ≥18 years at time of informed consent signature;
3. Histological confirmed locally advanced (any T N2-3) or metastatic urothelial bladder carcinoma, eligible to first-line treatment (previous neo adjuvant or adjuvant treatment must have been given and stopped more than one year before);
4. Evidence of progressive disease in the previous 6 months, documented by chest and/or abdominal CT-scan or MRI;
5. Measurable disease according to RECIST 1.1;
6. Karnofsky index ≥ 70%;
7. Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumour specimen (infiltrative urothelial bladder carcinoma or metastasis) collected within 12 months before Cycle 1 Day 1;
8. At least 3 weeks since the end of prior local intravesical treatment (BCG-therapy or ametycine) with resolution of all treatment-related toxicity to grade ≤1 (NCI CTCAE 4.0);
9. Palliative local treatment is allowed if performed ≥ 2 weeks prior study entry for radiotherapy, cimentoplasty or minor surgery, and ≥4 weeks for major surgery;
10. Adequate organ function as defined by the following criteria:

    1. Absolute White Blood Cells count (WBC) ≥ 2000 cells/mm3
    2. Absolute Neutrophils count (ANC) ≥ 1500 cells/mm3
    3. Platelets ≥100 000 cells/mm3
    4. Hemoglobin ≥ 9.0 g/dL
    5. Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
    6. Calculated creatinine clearance ≥ 60 mL/min
11. Women of childbearing potential must have a negative serum βHCG or urine pregnancy test within 7 days prior to initiation of treatment; both sexually active females and males (and their female partners) patients must agree to use two methods of effective contraception one of them being a barrier method, or to abstain from sexual activity during the study, for at least 3 months after the last administration of study treatment;
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures;
13. Patient affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

1. Other prior first-line therapy;
2. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment; focal radiation therapy less than 14 days prior to the first day of the first cycle;
3. Other invasive malignancy within 3 years (except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast); Patient with low risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 7 and PSA ≤ 10ng/mL) who are treatment-naïve and undergoing active surveillance are eligible;
4. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable;
5. Symptomatic central nervous system (CNS) metastases or untreated CNS metastases requiring concurrent treatment;
6. Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication;
7. Uncontrolled adrenal insufficiency;
8. Active chronic liver disease;
9. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
10. Active infection requiring systemic antibiotic;
11. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines;
12. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication);
13. Major surgery less than 28 days prior to the first day of the first cycle. Minor surgery less than 14 days prior to the first day of the first cycle;
14. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible;
15. History of primary immunodeficiency;
16. History of organ transplant including allogeneic stem-cell transplantation;
17. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3);
18. Women who are pregnant or lactating;
19. Known history of testing positive for HIV or known acquired immunodeficiency syndrome;
20. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Efficacy: objective response rate with RECIST 1.1 with GC + avelumab | At the end of cycle 6 (each cycle is 21 days)
Safety: proportion of severe toxicity with GC + avelumab | At the end of cycle 6 (each cycle is 21 days)

SECONDARY OUTCOMES:
Immunological capacities in peripheral blood of GC alone and GC+avelumab groups | During treatment and after the 6 cycles of treatment (EOT + 3, 6, 9 and 12 months
Specific immunological toxicity documented and recorded using NCI CTCAE version 4.0 | At the end of cycle 6 (each cycle is 21 days)
Duration of response | Up to 18 months
Progression-free survival | At 18 months in GC+avelumab treated patients
Overall survival | At 18 months in GC+avelumab treated patients
GC+avelumab efficacy according to the expression of PD-L1 at the tumor site | At the end of cycle 6 (each cycle is 21 days)
GC+avelumab efficacy according to the immune infiltrate populations at the tumor level and/or the tumor surroundings | At the end of cycle 6 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Alain RAVAUD, MD. PhD, Principal Investigator — University Hospital, Bordeaux
Locations (13):
- France (13):
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de cancérologie de l'Ouest - René Gauducheau, Nantes
  - Hôpital Européen Georges-Pompidou, AP-HP, Paris
  - Hôpital Saint-Louis, AP-HP, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gross-Goupil M, Domblides C, Lefort F, Ravaud A. Open-label randomized multi-center phase 2 study: gemcitabine cisplatin plus avelumab or gemcitabine cisplatin as first-line treatment of patients with locally advanced or metastatic urothelial bladder carcinoma: GCisAve. Bull Cancer. 2020 Jun;107(5S):eS1-eS7. doi: 10.1016/S0007-4551(20)30280-0. PMID 32620210